CLINICAL TRIAL: NCT02376725
Title: A Randomized Clinical Trial Comparing Phacoemulsification and Goniosynechialysis With Phacoemulsification Alone in the Management of Primary Angle Closure
Brief Title: Comparing Phaco/IOL Versus Phaco/IOL + Goniosynechialysis in Subjects With PACG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Rahat Husain, Consultant Ophthalmologist, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R796/80/2010
Record Dates: First submitted 2015-02-12; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Glaucoma, Angle-closure
Keywords: Goniosynechialysis
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phaco/IOL (Active Comparator): Cataract extraction using phacoemulsification technique with intraocular lens implant
  Interventions: Procedure: Phaco/IOL
- Phaco/IOL + goniosynechialysis (Active Comparator): Cataract extraction using phacoemulsification technique with intraocular lens implant with goniosynechialysis
  Interventions: Procedure: Phaco/IOL + goniosynechialysis

INTERVENTIONS:
Procedure: Phaco/IOL — Phaco/IOL refers to extracapsular cataract extraction (using phacoemulsification) and intraocular lens implantation
  Arms: Phaco/IOL
Procedure: Phaco/IOL + goniosynechialysis — Phaco/IOL refers to extracapsular cataract ectraction (using phacoemulsification) and intraocular lens implantation. Goniosynechialysis refers to mechanical breaking of peripheral anterior synechiae using a spatula and goniolens to view the drainage angle structures.
  Arms: Phaco/IOL + goniosynechialysis

SUMMARY:
The purpose of this study is to determine if phacoemulsification with intraocular lens implant (phaco/IOL) alone or combined with goniosynechialysis is better at controlling intraocular pressure in subjects with primary angle closure.

DETAILED DESCRIPTION:
Study Background

Glaucoma is the worlds' leading cause of irreversible blindness with nearly 7 million bilaterally blind due to the disease, by some estimates, and as such, represents a disease with significant associated morbidity. Furthermore, as glaucoma is primarily a disease of old age, as the number of elderly people in the world continues to rise, the number of people with glaucoma blindness is likely to have increasing economic burden and public health costs.

Primary glaucoma is classified into 2 types, Primary Open Angle Glaucoma (POAG) and Primary Angle Closure Glaucoma (PACG). Classification depends on configuration of the anterior chamber drainage angle, specifically if it is open or if it shows evidence of closure. The proportions of people with POAG and PACG are approximately equal, with the latter disease more common in Asians and women. Although the result of both diseases is progressive cupping of the optic disc with corresponding visual fields loss, the mechanism by which this occurs is thought to be quite different in the two diseases. In POAG the mechanism is still to be established but in PACG it is thought that apposition of the peripheral iris to the drainage angle results in damage to the trabecular meshwork (TM) and the formation of peripheral anterior synaechiae (PAS) which act as a mechanical obstruction of aqueous outflow via the trabecular meshwork. This in turn results in raised intraocular pressure (IOP) and subsequent optic nerve damage. Apposition can occur in anatomically predisposed eyes, although a physiological dynamic element is likely to be involved also. Areas of the TM not obstructed by PAS are likely to retain some function, although it is not clear if this is at the same level as in normal subjects. The functioning of the TM posterior to the areas of PAS has also yet to be established and it is hope that this study will help to elucidate this matter.

Conventional initial management of PACG is to perform laser peripheral iridotomy (LPI) to allow flow of aqueous from the posterior chamber to the anterior chamber through the iatrogenically created iridotomy. This has two benefits - in those subjects where pupillary-block is thought to be the mechanism for angle closure, it can reduce the risks of an acute rise in IOP occurring (acute angle closure). In other subjects with PAC, LPI has been shown to increase the drainage angle and this has led to lowering of the IOP in some subjects. However, in a retrospective review of 65 subjects with PACG who had had LPI, after 5 years follow-up the vast majority required further interventions (medications and/or surgery) to lower the IOP. Furthermore, PAS formation has been show to still occur in the presence of a patent PI. Clearly, the current conventional management strategy for PAC/PACG is inadequate and likely to lead to further ocular morbidity.

The poor results of LPI in the long-term for subjects with PACG in terms of IOP control has led many clinicians to study the effect of cataract surgery on IOP control in these patients. It was thought that removing the lens would increase anterior chamber depth and increase the drainage angle and hence increase outflow. Cataract surgery does indeed seem to open the drainage angle and its effects on IOP control have been promising. However, opening of the drainage angle may be limited in subjects with significant PAS. This could compromise the IOP lowering effect of cataract surgery in this group of patients. In such cases, cataract surgery with mechanical breaking of PAS (i.e. goniosynechialysis) might lower IOP to a greater extent than cataract surgery alone. Phacoemulsification + intraocular lens + Goniosynechialysis (PEI-GSL) has been carried out in several published studies, with all studies reporting a reduction in post-operative IOP compared to pre-operative. The main complications associated with PEI-GSL are excessive post-operative anterior chamber fibrinous reaction and anterior chamber bleeding. Theoretically, excessive pressure to break PAS could also cause iridodialysis or cyclodialysis, with resultant ocular hypotony. In an effort to reduce these complication risks, Varma and Fraser described phacoemulsification + intraocular lens + viscogonioplasty (PEI-VGP) in which a viscoelastic is used to break PAS in a non-iris contact method, rather than using an instrument to push the iris back. The authors proposed that this procedure would reduce the complications of PEI-GSL but still open the angle sufficiently. It is not clear however, if PEI-VGP would provide sufficient force to open areas of PAS and therefore be as efficacious as PEI-GSL in lowering IOP. Furthermore, there is no evidence that either PEI-GSL or PEI-VGP are superior to phacoemulsification + intraocular lens (PEI) alone in reducing IOP. Most surgeons will perform cataract surgery in patients with PAC/PACG and uncontrolled IOP. By adding the relatively simple step of goniosynechialysis during the surgical procedure, it has been proposed that this will result in further IOP lowering and hence less risk of glaucoma development/progression. This has yet to be proven.

An alternative treatment modality in subjects with PAC/PACG, visually significant cataract and high IOP, would be to perform phaco-trabeculectomy. Two recent randomized controlled trials published by Tham and co-workers, compared PEI versus phaco-IOL-trabeculectomy in subjects with medically controlled and medically uncontrolled angle-closure glaucoma. For the medically controlled group, there was no clinically significant difference in IOP lowering effect between the two surgical modalities. For the medically uncontrolled group, both modalities reduced IOP but the phaco-IOL-trabeculectomy group had a significantly lower IOP. However, the phaco-IOL-trabeculectomy group in both studies had a significantly higher complication rate than did the PEI group. Furthermore, only 4/27 (14.8%) of eyes in the PEI group (in the medically uncontrolled IOP study) required subsequent trabeculectomy to control IOP over the 2 years follow up period. In all these 4 cases, trabeculectomy was carried out successfully. Extrapolating from these data it would appear that although phaco-trabeculectomy does lower IOP more than PEI in patients with medically uncontrolled angle-closure glaucoma, many of these patients would not require 2 combined simultaneous procedures. Furthermore, trabeculectomy surgery has significant complication rates, even many years after the surgery is performed. Performing either PEI, or PEI-GSL (with or without viscoelastic assistance) would likely result in a significant reduction in IOP and still leave open the option of trabeculectomy (or glaucoma drainage device surgery) later on as the conjunctiva and sclera would be untouched. This multicentre study is designed to determine which of these 2 surgical options would superior in terms of efficacy and complications.

There have been no randomized controlled trials comparing PEI versus PEI-GSL (or PEI-VGP). There have been several case series and these will be summarized below.

Effect of phacoemulsification + intraocular lens on intraocular pressure in subjects with primary angle closure In patients with PAC or PACG, there is considerable evidence that PEI lowers IOP. Hayashi and coworkers, in a prospective study of 77 eyes of 77 consecutive patient with PACG found that IOP decreased significantly from baseline by an average of 6.1 ± 3.9 mmHg at 1 year follow up.5 Tham and co-workers showed an even more considerable decrease in IOP from a pre-operative mean of 24.4 mmHg to a mean of 15.4 mmHg at 15 months in a cohort of 27 patients with medically uncontrolled PACG.13 The same group examined the effect of PEI in a cohort of 35 eyes with medically controlled PACG.14 Pooling the results from both studies, PEI significantly reduced IOP from a pre-operative mean of 20.4 ± 5.8 mmHg to a mean of 14.6 ± 2.9 mmHg at 1 year, irrespective of pre-operative IOP control.

Effect of phacoemulsification + intraocular lens + goniosynechialysis on intraocular pressure in subjects with primary angle closure The largest case series on this topic, and the only prospective study performed on PEI-GSL was that performed by Teekhasaenee and coworkers. Fifty-two eyes of 48 patients (from Thailand) with PACG all underwent laser peripheral iridotomy but continued to have raised IOP defined as IOP >21 mmHg. Subjects underwent PEI-GSL and IOP decreased from a pre-operative mean of 29.7 ± 7.9 mmHg to 13.2 ± 2.9 mmHg at final examination (mean follow up 20.8 ± 15.5 months, range 5-76 months). This is a mean decrease of 16.5 mmHg.

There are 2 studies on the effect of PEI-VGP on IOP control, both retrospective case series. In the first, a consecutive series of 15 eyes of patients with refractory PACG, PEI-VGP reduced IOP significantly from 27.4 mmHg (on medication) to 14.1 mmHg (off all medication in 14/15 eyes), at 6 months.13 This represents a decrease of 13.3 mmHg. A subsequent study of 11 patients (11 eyes) on subjects with PACG (all of whom had refractory control despite patent peripheral iridotomy) showed a decrease in IOP from 39.4 mmHg pre-operatively to a mean of 13.4 mmHg after PEI-VGP at 7.8 months follow up.

Effect of phacoemulsification + intraocular lens alone or phacoemulsification + intraocular lens + goniosynechialysis on angle opening in subjects with primary angle closure

There are several studies which have shown that the drainage angle opens significantly after PEI in subjects with PAC/G.17;18 Only one paper described the effects of PEI on extent of peripheral anterior synaechiae. This showed that in subjects with PACG and PAS, there was a significant reduction in the extent of PAS after PEI, by approximately 25%.8 Most studies of PEI-GSL also describe opening of the drainage angle in subjects with PAC/G. Several studies also describe reduction in extent of PAS, including complete elimination of PAS.

The population to be studied will be all patients attending Singapore national Eye Centre (SNEC), Tan Tock Sen Hospital (TTSH), National University Hospital Singapore (NUHS), Vietnam National Institute of Ophthalmology, Thailand Faculty of Medicine Siriraj Hospital, Mahidol University and Hongkong, Queen Mary Hospital

This study will be conducted in compliance with the protocol, Singapore Good Clinical Practice (SGCP) and the applicable regulatory requirement(s).

Study Objectives and Purpose

To evaluate and compare the effect of two different surgical interventions in patients with primary angle-closure (with or without glaucoma), high intraocular pressure, and cataract.

These interventions are:

1. phacoemulsification + intraocular lens (PEI)
2. phacoemulsification + intraocular lens + goniosynechialysis (PEI-GSL).

Study Design

Experimental design This is prospective, longitudinal multicentre randomized control trial. The study sites will be SNEC, TTSH, NUHS, Vietnam National Institute of Ophthalmology, Thailand Faculty of Medicine Siriraj Hospital, Mahidol University and Hongkong, Queen Mary Hospital All subjects will undergo baseline and subsequent follow-up and evaluation in a standardized manner. Those who complete the informed consent process will be randomized to undergo either treatment with PEI or PEI-GSL. Subjects will then be followed-up for 12 months.

Study hypothesis We hypothesize that, compared to PEI, PEI-GSL will result in significantly lower IOP reduction both in the short and long term, with a reduction in amount of PAS, a wider drainage angle and a similar complication rate as PEI.

Patient Selection All subjects attending the glaucoma clinic at SNEC, TTSH, NUHS, Vietnam National Institute of Ophthalmology,Thailand Faculty of Medicine Siriraj Hospital, Mahidol University and Hongkong, Queen Mary Hospital will be eligible to be included in the study if they fulfill the inclusion/exclusion criteria (see below).

Once these criteria are fulfilled, subjects will be enrolled and divided into 2 groups using a random number generator. Group 1 will undergo PEI alone and Group 2 will undergo PEI-GSL.

Randomization and masking Block randomization method is used for randomization in this study. A pre-randomized list is generated according to Singapore Eye Research Institute's (SERI) standard operating procedure for randomization process by the clinic director and delegated stand-in. Following consent the study coordinator will contact the study centre (SERI) to obtain the randomization for each enrolled patient. Enrolled patient will be randomized to undergo either treatment with PEI or PEI-GSL. Randomization will be of patients and not eyes i.e. if two eyes of the same patient are eligible they will undergo the same intervention as allocated.

The investigator will be masked to the IOP measurement. Two individuals (an operator and a reader) will perform the IOP measurement. The operator operating the slit lamp and instrument dial will not be aware of the readings while the reader will read and record the results.

Surgical technique Anaesthetic will be general or peribulbar (approximately 3ml volume of 50/50 mix of 2% lignocaine and Marcaine with hyaluronidase). A superior or temporal clear corneal incision will be performed followed by creation of a paracentesis, injection of 3% sodium hyaluronate, 4% chondroitin sulfate (Viscoat, Alcon laboratories) and capsulorhexis. Hydrodissection is then performed using balanced salt solution and the lens is removed using phacoemulsification of the lens nucleus and aspiration (automated or manual) of cortical lens matter. After further injection of Viscoat, an acrylic injectable intraocular lens will be inserted into the capsular bag, its power having been determined pre-operatively based on biometric measurements. The Viscoat will then be removed (automated or manual), in the case of subjects undergoing PEI.

For those subjects PEI-GSL, the goniosynechialysis will be performed after partially filling the anterior segment with Sodium Hyaluronate 14mg/ml ("Healon GV", Advanced Medical Optics (AMO), California, USA). Using a goniolens (with coupling agent) to visualize those areas of PAS (defined pre-operatively), the viscoelastic will be used to break areas of PAS wherever possible, without touching the TM or iris. In cases where the viscoelastic is unable to break PAS, an iris repositor will be used to gently break the PAS in the areas where it exists. After this is performed, the surgery will continue as above, with removal of any remaining viscoelastic by automated or manual irrigation and aspiration.

Surgeries will be performed by senior ophthalmic surgeons. Any intraoperative complications (such as posterior capsular rupture, hyphaema, iris damage) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 30 years
2. Diagnosis of PAC or PACG. PAC is defined as previous documentation that the posterior trabecular meshwork was not visible for 180 degrees or more with gonioscopy (without indentation) previous to any LPI having been performed and evidence of appositional closure of the drainage angle by the peripheral iris, such as iris pigment in the angle or PAS, or any record of IOP > 21mmhg. PACG is defined as PAC as above and in addition glaucomatous optic neuropathy. Glaucomatous optic neuropathy is defined as functional and structural evidence of glaucomatous damage consistent with cup-disc ratio (CDR) 0.7 or asymmetry 0.2 between eyes or a neuroretinal rim width 0.1 CDR (at 11-10 or 5-7 0' clock). Glaucomatous field defect is diagnosed with reliable threshold visual field examination of the central 24-2 using Swedish Interactive Threshold Algoritm Standard (SITA-STD) 24-2 strategy, with glaucoma hemifield test results being outside normal limits, and with three or more non-edge contiguous points (except the horizontal nasal meridian) depressed to P<5%
3. IOP >21 mmHg or ≤ 21 mmHg on topical medication
4. More than or equal to 90 degrees of PAS (not necessarily contiguous)
5. Lens opacity deemed sufficient to be causing decreased vision in the opinion of the operating surgeon.
6. Informed consent

Exclusion Criteria:

1. Previous intraocular surgery (laser iridotomy is allowed)
2. Previous eye trauma resulting in documented damage to the drainage angle (such as angle recession)
3. For patients on warfarin, International Normalized ratio (INR) >3.0 on day of surgery
4. Evidence of moderate non-proliferative diabetic retinopathy, neovascularization, or rubeosis iridis
5. Chronic use of topical or systemic steroids
6. Any condition precluding or presumed to preclude reliable visual fields, disc stereo photography, or 12 months of follow up
7. Only eye (VA worse than 6/60 Snellen in non-study eye)
8. Advanced glaucoma with severe paracentral or generalized field deficit threatening fixation
9. Allergic to acetazolamide

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure as measured by Goldmann applanation tonometry | 1 year

SECONDARY OUTCOMES:
Per-operative and post-operative complications as determined by the examining/operating clinician | 1 year
Peripheral anterior synechiae development as measured by gonioscopy | 1 year
Degree of angle opening as measured by gonioscopy and anterior segment ocular coherence tomography | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye centre, Singapore, Singapore

REFERENCES:
- [Derived] Husain R, Do T, Lai J, Kitnarong N, Nongpiur ME, Perera SA, Ho CL, Lim SK, Aung T. Efficacy of Phacoemulsification Alone vs Phacoemulsification With Goniosynechialysis in Patients With Primary Angle-Closure Disease: A Randomized Clinical Trial. JAMA Ophthalmol. 2019 Oct 1;137(10):1107-1113. doi: 10.1001/jamaophthalmol.2019.2493. PMID 31294768